CLINICAL TRIAL: NCT03545516
Title: Randomized Control Trial for an Opioid Free Analgesic Pathway Post Cesarean Delivery
Brief Title: Wound Infiltration as Part of an Opioid Free Pain Management Pathway Following Cesarean Delivery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Richmond University Medical Center (Other)
Responsible Party: Principal Investigator, Nisha Lakhi, MD, Research Director, Richmond University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Post Cesarean Pain Management
Record Dates: First submitted 2018-03-22; First posted 2018-06-04 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative; Anesthesia, Local; Opioid Use
Keywords: Wound infiltration; Post Cesarean; Pain management; bupivacaine; dexmedetomidine; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Wound infiltration with a placebo
  Interventions: Drug: Placebo
- Bupivacaine (Experimental): Wound Infiltration with 20 mL (150mg) of 0.75% bupivacaine diluted with 5 mL of normal saline to give a 25 mL
  Interventions: Drug: Bupivacaine
- Bupivacaine and Dexmedetomidine (Experimental): Wound Infiltration with 20 mL (150mg) of 0.75% bupivacaine and 1.5 mcg/kg of dexmedetomidine will be diluted with normal saline to make 25 mL of solution .
  Interventions: Drug: Bupivacaine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine — Injection of bupivacaine into the surgical incision prior to its closure.
  Other Names: Bupivacaine wound infiltration
  Arms: Bupivacaine; Bupivacaine and Dexmedetomidine
Drug: Dexmedetomidine — Injection of dexmedetomidine ( an adjuvant) into the surgical incision prior to its closure.
  Other Names: Dexmedetomidine wound infiltration
  Arms: Bupivacaine and Dexmedetomidine
Drug: Placebo — Injection of a placebo into the surgical wound
  Arms: Placebo

SUMMARY:
This study will investigate the effect of three types of wound infiltration on post Cesarean opioid analgesia consumption when used in conjunction with an opioid free postoperative analgesia pathway.

DETAILED DESCRIPTION:
The subjects that meet the inclusion criteria of the study will be randomized preoperatively into three arms following a 1:1:1 ratio. During the intraoperative course one of three combinations of wound infiltration will be administered to subjects prior to the closure of the surgical incision. Subjects in Group I will receive a placebo of normal saline. Subjects in Group II will receive bupivacaine alone. Subjects in Group III will receive both bupivacaine and dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* All scheduled Cesarean deliveries with intrathecal or epidural anesthesia

Exclusion Criteria:

* Emergency Cesarean deliveries
* Multifetal gestation
* Subjects <18 years old
* Subjects belonging to a vulnerable population (including subjects with a known opioid addiction, subjects with a history of mental illness and prisoners)
* Cesarean delivery with general anesthesia
* Known allergy or hypersensitivity to any of the study medications
* Subjects that can't comprehend the visual analog scale for quantitative pain assessment

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 540 (Estimated)
Dates: Start 2018-09-17 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Total number of opioid free Cesarean deliveries | 1 year
  Measure the number of Cesarean deliveries that did not require opioid analgesia during the postoperative course

SECONDARY OUTCOMES:
Time to first rescue analgesia | 0 hour post-cesarean to time rescue analgeisa is administered]
  Measure the time to first rescue analgesia from immediate post operative (0 hour) till when the rescue analgesia is administered
Total opioid consumption | 0-14 days
  Measure the subjects total opioid consumption for the total duration of the postoperative course.
Side effects/Adverse reactions | 0-14 days
  Measure any side effects/allergic reactions attributed to use of any of the study drugs.
Postoperative hospital stay | 0-14days
  Measure the length of the post-operative hospital stay .
Complications from procedures | 0-14 days
  Measure any complications associated with the wound infiltration procedure
Breast feeding capacity | 0-14 days
  Assess the subject's capacity to breast feed during the postoperative course

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Lakhi, MD, Principal Investigator — Richmond University Medical Center
Locations (1):
- Richmond University Medical Center, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No